CLINICAL TRIAL: NCT03085212
Title: Strategies for Pregnancy Achievement (SPA): a Pilot Study
Brief Title: Strategies for Pregnancy Achievement
Acronym: SPA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Courtney D.Lynch, PhD MPH (Other)
Collaborators: The Cleveland Clinic (Other); University of California, Irvine (Other)
Responsible Party: Sponsor-Investigator, Courtney D.Lynch, PhD MPH, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015H0395
Record Dates: First submitted 2017-03-09; First posted 2017-03-21 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Fertility Disorders; Psychological Stress; Infertility; Infertility, Female
MeSH Terms: conditions — Stress, Psychological; Infertility; Infertility, Female

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online stress management program (Experimental): Participants will receive free access to Stress Free Now, which is an online stress management program developed by the Cleveland Clinic that uses mindfulness and cognitive-behavior therapy to help individuals learn to manage their stress.
  Interventions: Behavioral: Stress Free Now
- Wait list control (Active Comparator): Participants in this arm will receive free access to the Stress Free Now program at the end of the study.
  Interventions: Behavioral: Stress Free Now

INTERVENTIONS:
Behavioral: Stress Free Now — Online stress management program developed by the Cleveland Clinic that uses mindfulness and cognitive-behavioral therapy to help individuals manage their stress.

SUMMARY:
The purpose of pilot study application is to build on the investigators' previous work that established the prospective association between stress and infertility. Specifically, the investigators hope to collect the preliminary data necessary to make them competitive to submit a R01 application to NIH for funding of a full-scale randomized controlled trial of an internet-based stress management program to examine its efficacy in decreasing stress and increasing pregnancy rates among women who have tried to get pregnant for 6-12 months without success. The program called Stress Free Now (SFN) was developed at the Cleveland Clinic and has been shown to be effective in lowering stress in a variety of populations. The program introduces concepts of mindfulness and cognitive-behavioral therapy to assist individuals in managing their stress levels. The intervention includes Internet-based interaction, daily emails and recommended relaxation practice of at least four days per week. Using targeted Facebook Ads and other recruitment modalities, the investigators will randomize 40 women ages 18-34 who have been trying to conceive for 6-12 months without success. The PI has been enrolling women in a similar study using this mechanism and has found it to be an efficient and cost-effective method of identifying potentially eligible individuals. Women will be randomized to SFN or a wait list control condition and will be followed for up to three months post-randomization with weekly journals as they try to conceive. The primary outcome of this randomized controlled trial is stress level, as measured by salivary alpha-amylase, while the secondary outcome will be pregnancy rate at the end of the three-month follow-up period.

DETAILED DESCRIPTION:
To allow us to address the significant data gap regarding the efficacy of interventions to reduce stress and increase fecundity, we will conduct a randomized controlled trial of a proven 6-week online stress management program called Stress Free Now (SFN). Women will be randomized to SFN or a wait list control condition (i.e., participants assigned to the control arm with be offered SFN at the end of the study, even if they are already pregnant).

Women will be followed for three months from the date of randomization as they continue to try to conceive. Women who report pursuing fertility treatment will be censored on the day they report initiating treatment.

Participants will be recruited primarily using targeted Facebook Ads, though other modalities will also be used like local ads, and ResearchMatch. The PI used Facebook for recruitment for a similar study and found it to be a very efficient method for identifying women who are currently trying to conceive. We will preferentially target women in the Midwest for this pilot study in order to keep shipping costs low.

For the proposed study, the Facebook Ad will direct participants to the study website where they can obtain more information and complete a preliminary screening questionnaire using a secure online form. The brief screening questionnaire will assess whether the potential participant meets the above-mentioned eligibility criteria and will ask individuals to complete the State-Trait Anxiety Inventory (STAI), Trait Form, the 10-item Center for Epidemiologic Studies Depression Scale Revised (CESDR-10), and the four-item Perceived Stress Scale. Women who score ≥ 34 on the STAI and/or ≥ 10 on the CESDR-10 will be contacted by study staff and offered enrollment. These two assessments were chosen because they are the two instruments shown in the PI's prior work to correlate with salivary alpha-amylase level, which the biomarker that the PI has found to be associated with reduced fecundity.

Eligible women who complete the questionnaire and are found to be eligible will be informed via email and their address will be requested so that we can mail them an informed consent and HIPAA documents. The forms will be mailed and participants will be asked to return it to study staff using the prepaid envelope. When the signed forms are received, participants will be sent an email with a link to their baseline questionnaire. Once the baseline questionnaire has been completed, women will be sent their first saliva collection kit as well as five pregnancy tests for use during the study. If a woman reports on the baseline questionnaire that she is currently receiving infertility treatment, she will be exited from the study. In addition to collecting their saliva specimen (described below), women will be asked to use one of the enclosed pregnancy tests immediately, to record the results (i.e., pregnant or not pregnant), and to return the form with the saliva specimen. Any woman who reports that she is pregnant at baseline will be thanked and exited from the study.

Women who remain eligible will be randomized in a 1:1 ratio to the SFN intervention or waitlist control condition. The randomization scheme will be prepared and overseen by the study biostatistician. Women will be informed of their randomization status via email. For women randomized to the intervention, we will email staff at the Cleveland Clinic the woman's study identification number, name, email address, and phone number so that she can be given immediate access to Stress Free Now. For women randomized to the waitlist control condition, Cleveland Clinic staff will be sent her information at the end of the study (women who are randomized to the intervention group will receive access to Stress Free Now when they are done participating). During the data collection phase of the project all investigators will remain blinded to participants' randomization status except for the administrative support staff who will manage correspondence and mail the packages.

The intervention for this study will be a multifaceted online stress reduction program developed by the Cleveland Clinic. Each week for six weeks participants will be introduced to a new lesson. The topics include: being, being aware, being neutral, being you, being connected, and being joyful. The week will begin with a lesson guide recording that provides an overview of the lesson, then participants will be guided to read the short daily reading on the website (approximately one page) at which point they will be directed to complete the daily 20-25 minute relaxation practice, which is a recorded meditation or guided imagery exercise. The relaxation practices change with each week's lesson and participants will be directed to complete the relaxation practice at least four times a week. The relaxation practice recordings can be accessed at any time on the Stress Free Now website. Participants will receive daily emails with an inspirational quote that includes reminders to log in to do the day's reading and complete the daily relaxation practice. The daily readings discuss topics like stress, the importance of living in the present, perfectionism, optimism, mood, yoga, healthy eating, better sleep, loneliness and other related areas. Those data along with the number of times that the participant logged in to the Stress Free Now website will be recorded in the Cleveland Clinic's database and merged by participant ID with the rest of the study data. Women assigned to the control group will be given access to the intervention immediately upon completing the study (i.e., to fulfill the wait list control condition). It should be noted that while intervention crossover is always a concern, SFN has not been widely used to date (<50 public users last year) despite its demonstrated promise for reducing stress.

Our primary endpoint will be salivary alpha-amylase level, consistent with our prior work in this area. A highly experienced laboratory will quantify salivary cortisol and alpha-amylase as biomarkers of stress. Cortisol (micrograms/dL) will be measured using a highly sensitive enzyme immunoassay. Salivary alpha-amylase (U/mL) will be quantified using a commercially available kinetic reaction assay. Our secondary outcome will be pregnancy rate after three months of follow-up. Women will be asked to continue to participate in the study for the full three months, even if they become pregnant (this will allow us to assess levels of stress over time).

When sent their first saliva collection kit, participants will be provided detailed collection instructions, which will ask the participant to collect her first saliva sample the next morning within 10 minutes of awakening before eating, drinking, smoking, or brushing her teeth. Participants will be advised to freeze the collected sample in her home freezer for at least 12 hours prior to returning the sample to The Ohio State University using the provided prepaid insulated shipping container containing the frozen cold pack (see saliva collection form). In instances where women collects her sample too late (i.e., >30 minutes after awakening) or the sample arrives damaged or otherwise unusable, women will be asked to provide a replacement sample.

The Monday following randomization, women will be sent an email with a link to their first weekly journal. Specifically, women will be asked to record their answers to the journal questions in reference to days of bleeding, acts of intercourse, receipt of infertility treatment, pregnancy test results, health behaviors, stress level, and efforts to reduce stress. At weeks 6 and 12, women will also be asked to complete the PSS-4, the STAI-S Short Form, and the CESDR-10. Women will be asked to complete this journal at the end of each week (Mondays) until the end of the three-month follow-up period (12 journals total) or pregnancy, whichever comes first. Women who are randomized to the intervention will be sent a welcome email with their SFN username and password.

After 6 weeks of follow-up (corresponding to the end of the intervention for the group randomized to SFN), women will be mailed a second package containing saliva collection materials and will be asked to collect a second sample. Procedures will be identical to the first sample collection.

Study staff will maintain close contact with study participants to limit loss to follow-up. Participants in this randomized controlled trial will receive a $40 Amazon.com gift card for completing the study. As described above, women will also receive five digital pregnancy tests for use during the study; this will likely be viewed as a benefit by participants, but will also serve to increase the validity of the measurement of our primary endpoint. Upon exiting the study, all women will be asked to complete the study's exit form.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 18-34 years
* In a stable relationship with a male partner
* Has regular internet access
* Trying to get pregnant and last used contraception 6-12 months ago
* STAI-T score>=34 OR CESR-10 score >=10.

Exclusion Criteria:

* Currently pregnant
* Participant had a DepoProvera injection in the prior 12 months
* Currently receiving infertility treatment

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As we are studying the effect of stress reduction on pregnancy rate, participants must be female.
Enrollment: 40 (Estimated)
Dates: Start 2017-05-21 (Actual); Primary Completion 2019-04-03 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Stress level as measured by salivary alpha-amylase | Six weeks post randomization
  A salivary specimen will be collected to measure salivary alpha-amylase

SECONDARY OUTCOMES:
Pregnancy rate | Twelve weeks post randomization
  Rate of pregnancy as measured by study-provided home pregnancy test

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Lynch, PhD, Principal Investigator — The Ohio State University College of Medicine
Locations (1):
- The Ohio State University College of Medicine, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — https://www.facebook.com/spastudy2/